CLINICAL TRIAL: NCT00817323
Title: What is the Antidepressant Mechanism of Action of Quetiapine in Bipolar Depression? Evidence From Selective Neurotransmitter Depletion Studies
Brief Title: What is the Antidepressant Mechanism of Action of Quetiapine in Bipolar Depression?
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment did not take place for this research due to several delays and then one of the PIs moved out of the country and the project was closed
Sponsor: University of British Columbia (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: H07-02995
Record Dates: First submitted 2009-01-02; First posted 2009-01-06 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Bipolar Depression
Keywords: bipolar depression; atypical antipsychotic; remission; depletion; mood
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Quetiapine fumurate (Seroquel) (Experimental): See Detailed description
  Interventions: Procedure: Dietary amino-acid depletion

INTERVENTIONS:
Procedure: Dietary amino-acid depletion — See detailed description

SUMMARY:
PURPOSE The purpose of this study is to elucidate whether quetiapine fumurate (Seroquel) exerts its antidepressant activity in bipolar disorder through altering either serotonergic or catecholinergic activity.

HYPOTHESIS By depleting either serotonin or catecholamines in successfully treated bipolar patients, relapse will be induced and reveal which neurotransmitters are effected when receiving normal treatment

JUSTIFICATION While the exact mechanism of action of the classical antidepressants is not fully understood, strong evidence implicating serotonin and noradrenalin to be necessary (albeit insufficient) for the resolution of depression comes from neurotransmitter depletion studies. This biological evidence for each of these two neurotransmitters come from study paradigms in which the neurotransmitter (or its precursor) are selectively and effectively depleted from patients who have responded to antidepressants which either work through enhancing serotonin (for example, SRI antidepressants) or catecholamines (such as secondary amine tricyclics, Reboxetine, etc.). It has been shown, and replicated, that patients that respond to serotonin enhancing drugs precipitously and dramatically relapse when given a diet (often in the form of a milkshake) which is void of tryptophan, the precursor of serotonin. This diet often contains other long-chain amino acids to prevent any residual tryptophan in the system from entering the CNS. These patients who have then relapsed on the tryptophan-free diet have their tryptophan repleted and their mood improves often over a very short time frame (for example, five hours). When this technique is performed on patients responding to catecholamine-enhancing drugs there is no significant clinical effect. A similar approach can be taken with patients who respond to noradrelanine-enhancing drugs. Specifically, their catecholamine stores can be depleted by using dietary tyrosine. This reduces the synthesis of catecholamines and dopamine thus depleting pre-synaptic noradrenaline. For patients who responded to noradrenaline-enhancing drugs, this results in a relapse in terms of depressive symptomatology. When this dietary tyrosine strategy is applied to serotonin responders, there is no significant clinical effect.

DETAILED DESCRIPTION:
The study would be conducted at a single site: the University of British Columbia. This study would involve the recruitment of out-patient responders to quetiapine who previously had the diagnosis of bipolar disorder, depressed phase. These patients could then be randomized to receive either serotonergic or catecholinergic depletion, through tryptophan or tyrosine depletion respectively.

Baseline assessments would be conducted prior to the subjects being entered into the active phase of depletion. As the depletion phase is short, i.e. a number of days, this phase of the trial would be relatively short (i.e. one week).

Participants will see a clinician at a pre-depletion screening visit that occurs (maximum) 7 days prior to commencing depletion. In addition the a physical examination and taking medical history, inclusion/exclusion criteria will be verified, an ECG will be taken by a hospital cardiologist, and blood and urine samples will be collected for standard haematology/urinalysis, and a baseline assessment of amino acid and neurotransmitter levels. Patients would be maintained on their original dose of Quetiapine throughout the course of the study.

Amino acid and neurotransmitter concentrations will be determined on-site, by means of HPLC.

All depletion drinks will be mixed with 300ml of juice, to cover the taste of the amino acid mixture prepared. Male participants receiving a tyrosine-free formula, will drink a mixture of amino acids as administered in work by Sheenan et al (1996): L-isoleucine (7.5g); L-leucine (11.25g), L-lysine monohydrochloride (8.75g), L-methionine (2.5g), L-valine (8.75g), L-threonine (5g); L-tryptophan (1.25g). Female subjects will receive drinks of the same composition, but 20% less by weight of each amino acid. Similarly, the tryptophan-free formula for males will be as prepared by Hughes et al (2000, (Hughes, Dunne & Young 2000)), and formula that is 20% less, by weight, of amino acids will be used for females: L-alanine (5.5g); L-arginine (4.9g); L-cysteine (2.7g); L-glycine (3.2g); L-histidine 3.2g); L-isoleucine (8g); L-leucine (13.5); L-lysine monohydrochloride (11g); L-methionine (3g); L-phenylalanine (5.7g); L-proline (12.2g); L-serine (6.9g); L-threonine (6.5g); L-tyrosine (6.9g); L-valine (8.9g).

The depletion and post-depletion monitoring will occur daily for five (5) days, so depletion will begin on a Monday, unless circumstances require otherwise. Participants will be instructed to have a low-protein diet in the day prior to their second visit (total content of less than 20g), and fast from midnight until their visit. Subjects will arrive at the clinic at 9AM on day 1 and commence depletion, under the supervision of the screening physician, who will monitor the subject over the next four days, including at 0- and 4-hours post-depletion. At 24 hours post-depletion, a blood sample will be drawn for analysis of amino acid and neurotransmitter levels (5mL). Subjects will not be hospitalized during their participation, unless it is deemed necessary by clinician's judgment, but will be given 24-hour contact information for the attending physician. The same physician will see a given subject for the duration of their participation, and all raters involved in this study will have previously demonstrated an inter-rater reliability of 0.85 for all scales. At all visits (1-5), subjects will have mood assessed using a Visual Analog Scale, for self-rating, and by the Hamilton Rating-Scale for Depression. Concomitant medications will also be recorded.

At the final visit (96-hours post-depletion), a follow-up physical examination will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent
2. A diagnosis of Bipolar Disorder, depressed phase by Diagnostic and Statistical Manual of Mental Disorders- Fourth Edition (DSM-IV)
3. Females or males aged 19 to 65 years.
4. Female patients of childbearing potential must be using a reliable method of contraception and have a negative urine human chorionic gonadotropin (HCG) test at enrolment, and be in follicular phase of menstrual cycle for duration of depletion portion of study.
5. Able to understand and comply with the requirements of the study
6. Presently taking therapeutic doses of Quetiapine
7. In remission, as determined by attending clinician by scoring 7 or less on the HAM-D (17-item) at time of screening.

Exclusion Criteria:

1. Pregnancy or lactation
2. Any DSM-IV Axis I disorder not defined in the inclusion criteria
3. Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
4. Known intolerance or lack of response to quetiapine fumarate, as judged by the investigator
5. Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrolment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir
6. Use of any of the following cytochrome P450 inducers in the 14 days preceding enrolment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids
7. Administration of a depot antipsychotic injection within one dosing interval (for the depot) before randomisation
8. Substance or alcohol dependence at enrolment (including caffeine and nicotine dependence; except dependence in full remission), as defined by DSM-IV criteria
9. Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse by DSM-IV criteria within 6 months prior to enrolment
10. Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment
11. Unstable or inadequately treated medical illness (e.g. congestive heart failure, angina pectoris, hypertension) as judged by the investigator
12. Involvement in the planning and conduct of the study
13. Previous enrolment or randomisation of treatment in the present study.
14. Participation in another drug trial within 4 weeks prior enrolment into this study or longer in accordance with local requirements
15. A patient with Diabetes Mellitus (DM) fulfilling one of the following criteria:

    * Unstable DM defined as enrolment glycosylated hemoglobin (HbA1c) >8.5%.
    * Admitted to hospital for treatment of DM or DM related illness in past 12 weeks.
    * Not under physician care for DM
    * Physician responsible for patient's DM care has not indicated that patient's DM is controlled.
    * Physician responsible for patient's DM care has not approved patient's participation in the study
    * Has not been on the same dose of oral hypoglycaemic drug(s) and/or diet for the 4 weeks prior to randomisation. For thiazolidinediones (glitazones) this period should not be less than 8 Weeks.
    * Taking insulin whose daily dose on one occasion in the past 4 weeks has been more than 10% above or below their mean dose in the preceding 4 weeks Note: If a diabetic patient meets one of these criteria, the patient is to be excluded even if the treating physician believes that the patient is stable and can participate in the study.
16. An absolute neutrophil count (ANC) of 1.5 x 109 per liter
17. Currently taking any other antipsychotic, aside from Quetiapine.
18. Currently taking any antidepressant compounds, or in 8 weeks prior to enrolment.
19. Medical condition or known dietary sensitivity to depletion measures.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
To determine if a given depletion treatment induces relapse, measured as the mean HAM-D 17-item score of each group. A HAM-D score of 12 points or higher will be defined as relapse, measured 24-, 48- and 96-hours post-depletion. | 4 days

SECONDARY OUTCOMES:
Maximum change between each VAS item; change in HAM-D score; correlation of change in plasma tryptophan and catecholamine levels; correlation of change in plasma amino acid levels from baseline to 24 hours post-depletion. | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Alex Goumeniouk, Ph.D, Principal Investigator — University of British Columbia